CLINICAL TRIAL: NCT04592861
Title: A Prospective, Randomized, Phase 3 Trial of Carbon Ion Radiation Therapy Versus Standard Care for Locally Advanced Pancreatic Cancer
Brief Title: Carbon Ion RT for Locally Advanced Pancreatic Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study administratively closed out by the Einstein IRB. NO US enrolling sites.
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-11511
Record Dates: First submitted 2020-09-11; First posted 2020-10-19 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; carbon ion
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an open-label randomized trial. Subjects will be randomized in a 2:1 ratio to receive carbon ion radiotherapy versus standard care for locally advanced pancreatic cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Carbon ion radiotherapy (Experimental): Carbon ion radiotherapy will be administered 5 days each week (Monday-Friday). The prescription dose will be 60 GyE in 20 fractions, to be delivered over four weeks.
  Interventions: Radiation: carbon ion RT; Drug: Chemotherapy drug
- Routine standard of care (Active Comparator): Subjects on the control arm will not receive upfront radiotherapy but may receive radiotherapy (not carbon ion radiotherapy) if disease progression occurs.
  Interventions: Drug: Chemotherapy drug

INTERVENTIONS:
Radiation: carbon ion RT — daily carbon ion radiotherapy
  Arms: Carbon ion radiotherapy
Drug: Chemotherapy drug — Subjects who receive carbon ion radiotherapy may receive additional chemotherapy afterwards, at the discretion of the treating physicians. Subjects on the control arm are also expected to receive chemotherapy, using a regimen selected by the treating physicians.

SUMMARY:
This is an open-label randomized trial. Subjects will be randomized in a 2:1 ratio to receive carbon ion radiotherapy versus standard care for locally advanced pancreatic cancer. Subjects who receive carbon ion radiotherapy may receive additional chemotherapy afterwards, at the discretion of the treating physicians. Subjects on the control arm are also expected to receive chemotherapy, using a regimen selected by the treating physicians. Subjects on the control arm will not receive upfront radiotherapy but may receive radiotherapy (not carbon ion radiotherapy) if disease progression occurs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of adenocarcinoma of the pancreas
* Sum of maximum diameters of tumor and involved lymph nodes ≤6 cm T1-4N0-1M0,
* Unresectable disease by radiographic criteria (pancreas protocol CT or MRI) or surgical exploration within 30 days prior to registration, defined based on at least one of the following:

major venous thrombosis of the portal vein or SMV extending for several centimeters (precluding vein resection and reconstruction) encasement (>180°) of the SMA or proximal hepatic artery abutment of the celiac trunk

* No evidence of distant metastases, based upon axial (PET, CT, or MRI) imaging of the chest, abdomen, and pelvis within 30 days prior to registration
* ECOG Performance Status 0-1 within 30 days prior to registration
* Age ≥ 18
* CBC/differential obtained within 14 days prior to step 1 registration, with adequate bone marrow function defined as follows:
* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
* Platelets ≥ 100,000 cells/mm3
* Hemoglobin ≥ 9.0 g/dl (NOTE: The use of transfusion or other intervention to achieve Hgb ≥ 9.0 g/dl is acceptable)
* Additional laboratory studies within 14 days prior to registration demonstrating:

Creatinine < 2 mg/dl; GFR > 50 mL/min (Cockroft and Gault formula)

* Bilirubin < 1.5 x ULN
* ALT and AST ≤ 2.5 x ULN
* aPTT, PT ≤ 1.5 x ULN
* Patients must provide study specific informed consent prior to study entry.
* Women of childbearing potential and male participants must practice adequate contraception during protocol treatment and for at least 6 months following treatment For females of child-bearing potential, negative serum pregnancy test within 30 days prior to registration

Exclusion Criteria:

* More than one primary lesion
* Tumor invasion of the duodenum or stomach, confirmed by upper endoscopy
* Active malignancy, other than pancreatic cancer, for which systemic therapy is indicated. -History of adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy asides from hormonal therapy, adequately treated stage 1or 2 cancer currently in complete remission, or any other cancer that has been in complete remission for ≥ 5 years is permitted.
* Prior treatment for pancreatic cancer with surgical resection, external radiotherapy, or interstitial isotope implantation.
* Prior treatment for pancreatic cancer with a systemic therapy regimen/agent not included in the list below. Systemic therapy must be discontinued at least 14 days before study enrollment.
* FOLFIRINOX
* Gemcitabine/nab-paclitaxel
* Gemcitabine
* S-1
* Prior radiation therapy to the abdomen that would result in overlap of radiation therapy fields

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
Overall survival duration | The length of time from randomization until death from any cause for up to 24 months
  The length of time from randomization of treatment for cancer, that patients diagnosed with the disease are still alive.

SECONDARY OUTCOMES:
Progression-free survival duration | he length of time from study registration until disease progression at any site or death from any cause, up to 24 months
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse.
Local disease progression scored using RECIST 1.1 criteria | Up to 24 months
  A set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progress") during treatment
Adverse events as defined by CTCAE v5.0 | Up to 24 months
  A set of criteria for the standardized classification of adverse effects of drugs used in cancer therapy.
Quality-of-life, measured using the EORTC (European Organisation for Research and Treatment of Cancer) QLQ-C30 questionnaire | up to 24 months
  Questionnaire developed to measure the quality of life of cancer patients. Composite scores range from 0 to 100, with higher scores being more favorable.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Ohri, MD, Principal Investigator — Associate Professor
Locations (1):
- Shanghai Proton and Heavy Ion Center (SPHIC), Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No